CLINICAL TRIAL: NCT02201251
Title: A Randomized, Active-Controlled, Open-Label, Flexible-Dose Study to Assess the Safety and Tolerability of Topiramate as Monotherapy Compared With Levetiracetam as Monotherapy in Pediatric Subjects With New or Recent-Onset Epilepsy
Brief Title: A Study to Investigate the Safety of the Drugs Topiramate and Levetiracetam in Treating Children Recently Diagnosed With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CR104425; TOPMATEPY4067 (Other: Janssen Research & Development, LLC); 2012-001552-19 (EudraCT Number)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; Topiramate; Levetiracetam; Pediatric
MeSH Terms: conditions — Epilepsy | interventions — Topiramate; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Topiramate (Experimental): Topiramate weight based dosing for participants 2 to less than (<) 10 years of age not to exceed 350 mg/day (milligram per day), as tolerated; not to exceed 400 mg/day in participants 10-15 years of age, as tolerated.
  Interventions: Drug: Topiramate
- Levetiracetam (Active Comparator): Levetiracetam weight based dosing for all participants 2-15 years of age, not to exceed 60 milligram per kilogram per day (mg/kg/day), as tolerated. The maximum recommended daily dosage is 3,000 milligram (mg).
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Topiramate — Topiramate weight based dosing for participants 2 to <10 years of age not to exceed 350 mg/day, as tolerated; not to exceed 400 mg/day in participants 10-15 years of age, as tolerated.
  Arms: Topiramate
Drug: Levetiracetam — Levetiracetam weight based dosing for all participants 2-15 years of age, not to exceed 60 mg/kg/day, as tolerated. The maximum recommended daily dosage is 3,000 mg.
  Arms: Levetiracetam

SUMMARY:
The purpose of this study is to evaluate the safety of topiramate monotherapy compared with levetiracetam another standard antiepileptic drug (AED), as monotherapy for new-onset or recent-onset epilepsy (seizure disorder) on pediatric growth and maturation, bone mineralization, and kidney stone formation in children aged 2 to 15 years.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), open-label, multi-centric (conducted in more than one center) and 2-arm flexible-dose monotherapy study of topiramate compared with 1 another AED (levetiracetam) in pediatric participants with epilepsy. The total study duration will be up to of 1 year and 2 months per participant. The study consists of 3 parts: Screening (that is, up to 35 days before study commences on Day 1); Treatment (1 year) and post-treatment (30 days). Safety will primarily be evaluated by percentage of participants with kidney stones and change from baseline in bone mineral density at Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a clinical diagnosis of new-onset or recent-onset epilepsy characterized by partial-onset seizures (POS) (with or without secondary generalization) or primary generalized tonic-clonic seizures (PGTCS) in accordance with criteria of the International League Against Epilepsy. The epilepsy diagnosis must be within the previous 2 years before screening
* Caregivers (parents or legally acceptable representatives) of the participant must be able to accurately maintain the participant take-home record and seizure diary
* At screening, participant must have weight and height values within the 5th to 95th percentile for chronological age (based on standard Child Height and Weight Charts from the Centers for Disease Control [CDC])
* Participant must never have been treated for epilepsy (treatment-naïve) or have been treated with no more than 1 standard antiepileptic drug (AED) if temporary or urgent AED use was necessary. Previous AED exposure must not exceed either of the following: 1.)Thirty-one days immediately preceding enrollment, or 2.)A total of 6 months of previous AED exposure in the past if the AED has been discontinued for at least 1 year prior to enrollment
* Parents (or legally acceptable representatives) of the participant must sign an informed consent/permission document, indicating that they understand the purpose of and procedures required for the study and are willing to give permission for their child to participate in the study. Participant 7 years of age and older, capable of understanding the nature of the study, must provide assent for their participation

Exclusion Criteria:

* Participant has a surgically implanted and functioning vagus nerve stimulator
* Participant has a history of seizures as a result of a correctable medical condition, such as metabolic disturbance, toxic exposure, neoplasm, or active infection within 2 weeks prior to the first day of Screening
* Participant has had uncontrolled seizures while previously taking either topiramate or levetiracetam
* Participant has a history of non-epileptic seizures within 2 weeks prior to the first day of Screening
* Participant has myoclonic or absence seizures

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (41):
- United States (12):
  - Birmingham, Alabama
  - Los Angeles, California
  - Gulf Breeze, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Louisville, Kentucky
  - Columbus, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - San Antonio, Texas
  - Temple, Texas
- Argentina (2):
  - Buenos Aires
  - Córdoba
- Queensland, Australia
- Graz, Austria
- Belgium (2):
  - Leuven
  - Namur
- Saskatoon, Saskatchewan, Canada
- France (4):
  - Brest
  - Bron
  - Paris
  - Toulouse
- Germany (2):
  - München
  - Tübingen
- Hungary (4):
  - Balassagyarmat
  - Budapest
  - Debrecen
  - Veszprém
- Philippines (2):
  - Cebu
  - Manila
- Poland (3):
  - Krakow
  - Poznan
  - Warsaw
- Russia (2):
  - Saint Petersburg
  - Ulyanovsk
- Durban, South Africa
- Taiwan (4):
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: Participants received topiramate weight-based sprinkle capsule and tablet, as tolerated (not to exceed 350 milligrams per day [mg/day] for participants 2 to less than [<] 10 years of age, and not to exceed 400 mg/day for participants 10 to 15 years of age), twice daily (BID) for up to 1 year during open-label treatment phase. Participants were to either continue on commercially available topiramate or were tapered off of study drug over a period of up to 2 weeks during post-treatment phase of 30 days.
- Levetiracetam: Participants received levetiracetam weight-based tablet or oral solution, as tolerated (not to exceed 60 milligrams per kilogram per day [mg/kg/day] for participants 2 to 15 years of age). The daily dosage was increased every 2 weeks by increments of 20 mg/kg/day to the recommended daily dosage of 60 mg/kg/day. The maximum recommended daily dosage was 3000 mg (1500 mg BID) for up to 1 year during open-label treatment phase. Participants were to either continue on commercially available levetiracetam or were tapered off of study drug over a period of up to 2 weeks during post-treatment phase of 30 days.
Period: Overall Study
Arm/Group | Topiramate | Levetiracetam
Started | 28 | 35
Completed | 24 | 32
Not Completed | 4 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Noncompliance with Study Drug | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Levetiracetam | Total
Number analyzed (Participants) | 28 | 35 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (2.76) | 9.3 (3.29) | 9.6 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 12 | 17 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 10 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 25 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRIA | 0 | 2 | 2
  CANADA | 0 | 1 | 1
  HUNGARY | 4 | 5 | 9
  ITALY | 3 | 4 | 7
  PHILIPPINES | 1 | 2 | 3
  POLAND | 8 | 8 | 16
  RUSSIAN FEDERATION | 2 | 4 | 6
  TAIWAN | 9 | 8 | 17
  UNITED STATES | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight Z-score up to Month 1
Description: The Z-Score indicates how many standard deviations (SD) a participant has from the population normal values. The body weight z-scores were designed to take into account the amount of weight gain that was expected due to normal growth in children and adolescents. Body weight data were converted to Z-scores using the Statistical Analysis System (SAS) programs provided by the Centers for Disease Control (CDC) for the calculation of the 2000 CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 1 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 1
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 27 | 34
Z-score | -0.112 (0.1220) [lower limit 0.1220] | -0.014 (0.1244) [lower limit 0.1244]

2. Primary Outcome: Change From Baseline in Weight Z-score up to Month 3
Description: The Z-Score indicates how many SD a participant has from the population normal values. The body weight z-scores were designed to take into account the amount of weight gain that was expected due to normal growth in children and adolescents. Body weight data were converted to Z-scores using the SAS programs provided by the CDC for the calculation of the 2000 CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 3 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 27 | 34
Z-score | -0.201 (0.2094) [lower limit 0.2094] | -0.027 (0.1802) [lower limit 0.1802]

3. Primary Outcome: Change From Baseline in Weight Z-score up to Month 6
Description: The Z-Score indicates how many SD a participant has from the population normal values. The body weight z-scores were designed to take into account the amount of weight gain that was expected due to normal growth in children and adolescents. Body weight data were converted to Z-scores using the SAS programs provided by the CDC for the calculation of the 2000 CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 6 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 24 | 33
Z-score | -0.319 (0.2496) [lower limit 0.2496] | -0.070 (0.2304) [lower limit 0.2304]

4. Primary Outcome: Change From Baseline in Weight Z-score up to Month 9
Description: The Z-Score indicates how many SD a participant has from the population normal values. The body weight z-scores were designed to take into account the amount of weight gain that was expected due to normal growth in children and adolescents. Body weight data were converted to Z-scores using the SAS programs provided by the CDC for the calculation of the 2000 CDC growth charts. The mean (SD) change in Z scores from baseline up yo Month 9 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 24 | 32
Z-score | -0.326 (0.3235) [lower limit 0.3235] | -0.110 (0.3584) [lower limit 0.3584]

5. Primary Outcome: Change From Baseline in Weight Z-score up to Month 12
Description: The Z-Score indicates how many SD a participant has from the population normal values. The body weight z-scores were designed to take into account the amount of weight gain that was expected due to normal growth in children and adolescents. Body weight data were converted to Z-scores using the SAS programs provided by the CDC for the calculation of the 2000 CDC growth charts. The mean (SD) change in Z scores from baseline to Month 12 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 24 | 32
Z-score | -0.351 (0.3905) [lower limit 0.3905] | -0.065 (0.3026) [lower limit 0.3026]

6. Primary Outcome: Change From Baseline in Height Z-score up to Month 1
Description: Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from minus (-) 3 to plus (+) 3; 0 equal to (=) same mean, greater than (>) 0 a greater mean, and less than (<) 0 a lesser mean than the standard. Growth parameters were compared to a standard defined by CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 1 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 27 | 33
Z-score | 0.004 (0.0870) [lower limit 0.0870] | -0.015 (0.1017) [lower limit 0.1017]

7. Primary Outcome: Change From Baseline in Height Z-score up to Month 3
Description: Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from -3 to +3; 0 =same mean, >0 a greater mean, and <0 a lesser mean than the standard. Growth parameters were compared to a standard defined by CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 3 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 27 | 34
Z-score | -0.036 (0.1452) [lower limit 0.1452] | 0.017 (0.1631) [lower limit 0.1631]

8. Primary Outcome: Change From Baseline in Height Z-score up to Month 6
Description: Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from -3 to +3; 0 =same mean, >0 a greater mean, and <0 a lesser mean than the standard. Growth parameters were compared to a standard defined by CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 6 for the total safety population for all age cohorts combined were presented.
Time Frame: Baseline up to Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 24 | 33
Z-score | -0.008 (0.1753) [lower limit 0.1753] | 0.077 (0.2670) [lower limit 0.2670]

9. Primary Outcome: Change From Baseline in Height Z-score up to Month 9
Description: Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from -3 to +3; 0 =same mean, >0 a greater mean, and <0 a lesser mean than the standard. Growth parameters were compared to a standard defined by CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 9 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 24 | 32
Z-score | -0.059 (0.2337) [lower limit 0.2337] | 0.086 (0.2929) [lower limit 0.2929]

10. Primary Outcome: Change From Baseline in Height Z-score up to Month 12
Description: Z-Score was a statistical measure to evaluate how a single data point compares to a standard. It described whether a mean was above or below the standard and how unusual the measurement is with range from -3 to +3; 0 =same mean, >0 a greater mean, and <0 a lesser mean than the standard. Growth parameters were compared to a standard defined by CDC growth charts. The mean (SD) change in Z scores from baseline up to Month 12 for the total safety population for all age cohorts combined were presented. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean.
Time Frame: Baseline up to Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 24 | 32
Z-score | -0.057 (0.2734) [lower limit 0.2734] | 0.088 (0.3315) [lower limit 0.3315]

11. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) Z-score up to Month 6
Description: The BMD was measured by dual energy X-ray absorptiometry (DEXA) for the posterior-anterior lumbar spine (L1_L4) and total body less head area. The Z-Score is the number of standard deviations a participant's BMD differs from the average BMD of their age, sex and ethnicity. Positive scores indicate BMD above the mean; positive values are "best values" and negative values are "worst values". Positive changes from baseline indicated an improvement in condition.
Time Frame: Baseline up to Month 6
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies the number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies the number of participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 25 | 32
Z-score
  Lumbar spine: number analyzed (Participants) | 24 | 32
  Lumbar spine | -0.181 (0.2590) | 0.035 (0.2606)
  Total body less head: number analyzed (Participants) | 25 | 30
  Total body less head | -0.180 (0.2647) | 0.102 (0.2574)

12. Primary Outcome: Change From Baseline in BMD Z-score up to Month 12
Description: The BMD was measured by DEXA for the posterior-anterior lumbar spine (L1_L4) and total body less head area. The Z-Score is the number of standard deviations a participant's BMD differs from the average BMD of their age, sex and ethnicity. Positive scores indicate BMD above the mean; positive values are "best values" and negative values are "worst values". Positive changes from baseline indicated an improvement in condition.
Time Frame: Baseline up to Month 12
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug. Here 'N' (number of participants analyzed) signifies the number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies the number of participants evaluable at a specified category.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 24 | 30
Z-score
  Lumbar spine: number analyzed (Participants) | 23 | 30
  Lumbar spine | -0.346 (0.3461) | 0.084 (0.3552)
  Total body less head: number analyzed (Participants) | 24 | 28
  Total body less head | -0.367 (0.3170) | 0.054 (0.3766)

13. Primary Outcome: Change From Baseline in Bone Mineral Content (BMC)-Z Score up to Month 6
Description: The BMC is an estimate of the amount of mineral (such as calcium) in the bone, which was assessed by DEXA scan for the posterior-anterior lumbar spine (L1_L4) and total body less head area. Positive changes from baseline indicated an improvement in condition.
Time Frame: Baseline up to Month 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 15 | 19
Z-score
  Lumbar spine: number analyzed (Participants) | 14 | 19
  Lumbar spine | -0.141 (0.2155) | 0.075 (0.2806)
  Total body less head | -0.242 (0.2516) | 0.151 (0.2154)

14. Primary Outcome: Change From Baseline in BMC-Z Score up to Month 12
Description: as for outcome 13
Time Frame: Baseline up to Month 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 15 | 18
Z-score
  Lumbar spine: number analyzed (Participants) | 14 | 18
  Lumbar spine | -0.274 (0.3123) | 0.124 (0.3584)
  Total body less head | -0.266 (0.6800) | 0.017 (0.2533)

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. TEAE are defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.
Time Frame: Up to Day 390
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 28 | 35
Participants | 25 | 29

16. Secondary Outcome: Percentage of Participants With Kidney Stones
Description: Percentage of participants with kidney stones were reported.
Time Frame: Up to Day 390
Population: Safety analysis set included all randomized subjects who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate | Levetiracetam
Number analyzed (Participants) | 28 | 35
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 390
Description: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Topiramate | Levetiracetam
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/28 | 5/35
Other Adverse Events (participants affected / at risk) | 25/28 | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=28) | Levetiracetam (N=35)
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=28) | Levetiracetam (N=35)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Middle Ear Effusion (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Epigastric Discomfort (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Influenza Like Illness (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
Sluggishness (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Ear Infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Gastroenteritis Enteroviral (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 7
Pharyngitis (Infections and infestations) | 3 | 0
Pneumococcal Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pulpitis Dental (Infections and infestations) | 0 | 1
Respiratory Tract Infection Viral (Infections and infestations) | 1 | 3
Rhinitis (Infections and infestations) | 2 | 3
Scarlet Fever (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 3 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Staphylococcal Pharyngitis (Infections and infestations) | 0 | 1
Systemic Viral Infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 7
Varicella (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Lip Injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ammonia Decreased (Investigations) | 0 | 1
Blood Potassium Increased (Investigations) | 0 | 1
Blood Triglycerides Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Vitamin D Decreased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Balance Disorder (Nervous system disorders) | 0 | 1
Cognitive Disorder (Nervous system disorders) | 1 | 0
Disturbance in Attention (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dizziness Exertional (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 9
Hypoaesthesia (Nervous system disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 2
Mental Impairment (Nervous system disorders) | 1 | 0
Partial Seizures (Nervous system disorders) | 1 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 2 | 3
Affective Disorder (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 2 | 0
Emotional Disorder (Psychiatric disorders) | 0 | 1
Hyposomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 0 | 5
Learning Disorder (Psychiatric disorders) | 1 | 0
Mood Swings (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 2
Sleep Disorder (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to futility of enrollment, the enrollment was stopped early; however, all enrolled participants completed the full course of the trial excluding 7 participants (reasons captured in "participant flow"). Also, there was no exposure to topiramate in 2 to 5 years age cohort. Therefore, no conclusions can be made with regard to this age group due to the absence of comparability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT02201251/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT02201251/SAP_001.pdf